CLINICAL TRIAL: NCT06619964
Title: Developing Evidence to Inform Regulatory Policy on Nicotine Content in E-Liquids
Status: Enrolling by invitation | Type: Observational
Sponsor: Rochester Institute of Technology (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Rochester (Other)
Responsible Party: Principal Investigator, Risa Robinson, Professor, Rochester Institute of Technology
Other Study IDs: 1R01DA057687 (NIH); 1R01DA057687-01A1 (NIH)
Record Dates: First submitted 2024-09-28; First posted 2024-10-01 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Nicotine Addiction
Keywords: electronic cigarettes; nicotine addiction; eliquid nicotine concentration; perception of risk; health effects; biomarkers of exposure; subjective affect
MeSH Terms: conditions — Tobacco Use Disorder; Vaping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn if electronic cigarette users who currently choose to use lower nicotine eliquids have reduced harm compared those who choose higher nicotine eliquids.

The main questions it aims to answer are:

* Do lower nicotine users actually consume less nicotine compared to higher nicotine users?
* Do lower nicotine users have lower amounts of harmful and potentially harmful constituent exposures compared to higher nicotine users?
* Do lower nicotine users perceive their choice of product to be less harmful than higher nicotine products? Researchers will monitor ecig users of different nicotine concentrations for two weeks in their natural environment to determine how much eliquid and nicotine they consumed, assess their daily mood and craving, and measure exposure and health effect.

Participants will:

* Complete surveys on history of tobacco use, nicotine dependence and perception.
* Use their electronic cigarette with their usual nicotine eliquid ad lib for two weeks in their natural environment.
* Complete daily questionnaires for mood and craving for two weeks in their natural environment.
* Collect three salivary samples at home, morning, afternoon and evening, each day for two weeks, in their natural environment.
* Use a topography monitor to record puffing behavior for every puff taken during week two, in their natural environment.
* Provide saliva, urine and blood samples in the lab at the end of each week.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 yrs or older
* Pod-style or pen-style users, not adjustable for power or airflow, nicotine greater than 0 mg/mL
* Current everyday users
* Use history of at least 30 days
* No current use of combustible tobacco product, or nicotine replacement therapy
* CO less than 6 ppm at intake
* No plans to quit tobacco use in the next 30 days

Exclusion Criteria:

* History of acute or chronic asthma
* Previous diagnosis of cancer
* Other chronic medical conditions
* Use of chronic prescription medications
* Pneumonia in prior six weeks
* Upper respiratory tract infection or other febrile illness in previous 2 weeks
* On antioxidants or anti-inflammatory therapy
* Pregnant women or women who intend to become pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residence of the Greater Rochester, NY area
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean daily salivary cotinine | From enrollment to the end of observation at 2 weeks.
  Nicotine exposure as indicated by mean daily salivary cotinine will be compared for lower versus higher nicotine strength regular ecig users, on a continuous scale. This will determine the extent to which reduced nicotine products result in lower nicotine exposure.

CONTACTS AND LOCATIONS:
Locations (1):
- Rochester Institute of Technology, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided